CLINICAL TRIAL: NCT05952219
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-379 in Healthy Volunteers Under Fed Conditions
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of CKD-379
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A125_04BE2302
Record Dates: First submitted 2023-07-10; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: Reference drug(D759+D745+D029+D150) Period 2: Test drug(CKD-379)
  Interventions: Drug: CKD-379; Drug: D759+D745+D029+D150
- Sequence 2 (Experimental): Period 1: Test drug(CKD-379) Period 2: Reference drug(D759+D745+D029+D150)
  Interventions: Drug: CKD-379; Drug: D759+D745+D029+D150

INTERVENTIONS:
Drug: CKD-379 — 2 tablet administration under fed condition
Drug: D759+D745+D029+D150 — 4 tablet co-administration under fed condition

SUMMARY:
A study to compare the pharmacokinetics and safety between CKD-379 and D759, D745, D029, D150 combination

DETAILED DESCRIPTION:
A randomized, open-label, single dose, crossover study to evaluate the pharmacokinetic profiles and safety of CKD-379 in healthy volunteers under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Between 19 aged and 50 aged in healthy adult
* 18.0kg/m2≤body mass index(BMI)≤27.0kg/m2 and 50.0kg≤Body weight≤90.0kg

Exclusion Criteria:

* Have clinical significant medical history or disease that blood, kidney(moderate nephropathy and etc.), endocrine system(type I or type II diabetes mellitus, diabetic ketoacidosis, diabetic coma and etc.), respiratory system, gastrointestinal system, urinary system, cardiovascular system(heart failure, Torsades de pointes and etc.), liver(moderate liver disorder and etc.), mental system, nervous system, immune system
* Have a gastrointestinal disease(Crohn's disease, ulcer etc.) history that can effect drug absorption or surgery
* Those who are pregnant or breastfeeding
* Those who are deemed inappropriate to participate in clinical trial by investigators

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
AUCt | 0~48hours
  Maximum plasma concentration of the drug
Cmax | 0~48hours
  Area under the concentration-time curve from the time of dosing to the last measurable concentration

CONTACTS AND LOCATIONS:
Overall Officials: Seol Ju Moon, M.D, Ph.D., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea